CLINICAL TRIAL: NCT03713606
Title: Serum Biomarkers Associated With Endothelial Dysfunction and Immune Inflammation for Portal Hypertension in Cirrhosis (Pan-CHESS1802)
Brief Title: Serum Biomarkers for Portal Hypertension in Cirrhosis (Pan-CHESS1802)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Beijing YouAn Hospital (Other); Shandong Provincial Hospital (Other Government); Beijing Shijitan Hospital, Capital Medical University (Other); Beijing Friendship Hospital (Other); Xingtai People's Hospital (Other); Beijing 302 Hospital (Other)
Responsible Party: Principal Investigator, Xiaolong Qi, Director, Hepatic Hemodynamic Lab, Nanfang Hospital, Southern Medical University
Other Study IDs: Pan-CHESS1802
Record Dates: First submitted 2018-10-18; First posted 2018-10-22 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Hypertension, Portal
Keywords: Portal hypertension; serum biomarker; diagnosis
MeSH Terms: conditions — Hypertension, Portal; Disease | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Overall eligible participants: Eligible participants will receive HVPG measurement by catheterization of a hepatic vein with a balloon catheter and run blood tests.
  Interventions: Procedure: HVPG measurement

INTERVENTIONS:
Procedure: HVPG measurement — HVPG obtained by means of catheterization of a hepatic vein with a balloon catheter.
  Other Names: Blood test

SUMMARY:
This is a prospective, multi-center diagnostic trial conducted at 6 liver centers in China designed to study the correlation between serum biomarkers associated with endothelial dysfunction and immune inflammation and hepatic venous pressure gradient in cirrhosis.

DETAILED DESCRIPTION:
Hepatic venous pressure gradient (HVPG) is the gold standard for assessing portal pressure, of which the measurement is invasive and therefore not suitable for routine clinical practice. The detection of serum biomarkers is potential for noninvasive diagnosis of portal hypertension in cirrhosis. However, many are still in the exploratory phases of testing and are not yet ready to enter clinical practice. This study prospectively enrolled participants in 6 liver centers (Beijing YouAn Hospital, Shandong Provincial Hospital, Beijing Shijitan Hospital, Beijing Friendship Hospital, Xingtai People's Hospital, and 302 Hospital of PLA) in China designed to study the correlation between serum biomarkers associated with endothelial dysfunction and immune inflammation and HVPG in cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 years;
* confirmed cirrhosis based on histologic examination of liver or combined physical, laboratory, and radiologic findings, including a nodular surface, a coarse texture, and an enlarged caudate lobe of the liver.

Exclusion Criteria:

* prior drug therapy (e.g. β-blocker, vasopressin) within two weeks
* prior surgeries (e.g. TIPS, partial splenic embolization/ devascularization, splenectomy, liver transplantation)
* non-sinusoidal portal hypertension & HCC inability to adhere to study procedures
* pregnancy or unknown pregnancy status
* no informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cirrhotic portal hypertension
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2018-09-30 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between serum biomarkers and HVPG | 1 day
  Correlation between serum biomarkers and HVPG

SECONDARY OUTCOMES:
Correlation between serum biomarkers and HVPG in HBV subgroup | 1 day
  Correlation between serum biomarkers and HVPG in a subgroup of patients with HBV-related cirrhosis

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong Qi, M.D., Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (6):
- China (6):
  - 302 Hospital of PLA, Beijing
  - Beijing Friendship Hospital, Beijing
  - Beijing Shijitan Hospital, Beijing
  - Beijing YouAn Hospital, Beijing
  - Shandong Provincial Hospital, Jinan
  - Xingtai People's Hospital, Xingtai

IPD SHARING:
Plan to Share IPD: Undecided
Undecided.

REFERENCES:
- [Background] Groszmann RJ, Wongcharatrawee S. The hepatic venous pressure gradient: anything worth doing should be done right. Hepatology. 2004 Feb;39(2):280-2. doi: 10.1002/hep.20062. No abstract available. PMID 14767976
- [Background] Waidmann O, Brunner F, Herrmann E, Zeuzem S, Piiper A, Kronenberger B. Macrophage activation is a prognostic parameter for variceal bleeding and overall survival in patients with liver cirrhosis. J Hepatol. 2013 May;58(5):956-61. doi: 10.1016/j.jhep.2013.01.005. Epub 2013 Jan 16. PMID 23333526
- [Background] Buck M, Garcia-Tsao G, Groszmann RJ, Stalling C, Grace ND, Burroughs AK, Patch D, Matloff DS, Clopton P, Chojkier M. Novel inflammatory biomarkers of portal pressure in compensated cirrhosis patients. Hepatology. 2014 Mar;59(3):1052-9. doi: 10.1002/hep.26755. Epub 2014 Jan 29. PMID 24115225
- [Background] Ferlitsch M, Reiberger T, Hoke M, Salzl P, Schwengerer B, Ulbrich G, Payer BA, Trauner M, Peck-Radosavljevic M, Ferlitsch A. von Willebrand factor as new noninvasive predictor of portal hypertension, decompensation and mortality in patients with liver cirrhosis. Hepatology. 2012 Oct;56(4):1439-47. doi: 10.1002/hep.25806. Epub 2012 Aug 27. PMID 22532296
- [Background] Qi X, Berzigotti A, Cardenas A, Sarin SK. Emerging non-invasive approaches for diagnosis and monitoring of portal hypertension. Lancet Gastroenterol Hepatol. 2018 Oct;3(10):708-719. doi: 10.1016/S2468-1253(18)30232-2. PMID 30215362